CLINICAL TRIAL: NCT04667455
Title: Improving Care for Children With Congenital Heart Disease by Cardiovascular Biomarker Profiling and Advanced Non-invasive Cardiac Imaging Techniques.
Brief Title: Improving Care for Children With Congenital Heart Disease.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Region Jönköping County (Other Government); Göteborg University (Other)
Responsible Party: Principal Investigator, Henning Clausen, MD, Hennnig Clausen, MD, Lund University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019-05490
Record Dates: First submitted 2020-10-26; First posted 2020-12-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Heart Disease Congenital; Ventricular Septal Defect; Atrial Septal Defect; Patent Ductus Arteriosus; Partial Anomalous Pulmonary Venous Connection; Aortopulmonary Window; Cardiovascular Diseases
Keywords: congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Ventricular; Heart Septal Defects, Atrial; Ductus Arteriosus, Patent; Aortopulmonary Septal Defect; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: case-control cohort
Who Masked: Participant, Care Provider
Masking Description: Participant and standard clinical care providers will be blinded to biomarker analyses and advanced cardiac imaging findings throughout the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control subjects (No Intervention): Infants and Children with no evidence of congenital heart disease based on clinical examination and echocardiography / standard ECG assessment where necessary.
- Congenital heart disease subjects (Active Comparator): Infants and Children with evidence of predefined congenital heart disease lesions based on clinical examination, echocardiography and standard ECG assessment
  Interventions: Diagnostic Test: Biomarker analysis at enrolment; Diagnostic Test: Biomarker analyses throughout the study

INTERVENTIONS:
Diagnostic Test: Biomarker analysis at enrolment — Controls will be compared to cases using blood-based biomarker analyses and non-invasive cardiac imaging techniques to improve early diagnosis and risk stratification of cases
  Other Names: blood-based and non-invasive cardiac imaging modalities at enrolment
  Arms: Congenital heart disease subjects
Diagnostic Test: Biomarker analyses throughout the study — Controls will be compared to cases using blood-based biomarker analyses and non-invasive cardiac imaging techniques to improve early diagnosis and risk stratification of cases
  Other Names: blood-based and non-invasive cardiac imaging modalities throughout the study
  Arms: Congenital heart disease subjects

SUMMARY:
Establish a cardiovascular biomarker profile to help screening for congenital heart disease in infants and children as well as use non-invasive cardiac imaging in combination with such profiling to better predict the need for future cardiac interventions such as open heart surgery or cardiac catheter intervention in selected types of with congenital heart disease.

DETAILED DESCRIPTION:
Analysing circulating cardiovascular biomarkers using blood samples should improve identification of congenital heart disease in newborns, in particular for those needing future cardiac interventions.

Comparing such biomarker profiles and non-invasive cardiac imaging results over time in infants and children should lead to better understanding of the complex cardiovascular remodelling processes in common congenital heart lesions, such as atrial or ventricular septal defects. This in turn should lead to an improved risk factor assessment model to guide treatment decisions in children with congenital heart disease in the foreseeable future.

To test our hypothesis, that cardiovascular biomarker profiling and non-invasive cardiac imaging findings in infants and children with congenital heart disease, differs from healthy controls, we will assess controls at enrolment and follow cases with predefined congenital heart disease lesions over a maximum of three years or up till one year after open heart surgery / cardiac catheter intervention to correct such lesions.

Infants and children resident in designated healthcare regions of Sweden will be invited to participate after study advertisement. Written informed consent will be obtained from legal guardians and assent will be sought from children who can communicate verbally with the dedicated paediatric research team.

Healthy subjects 0-17 years at enrolment will undergo i.e. standard electrocardiogram (ECG), echocardiography and blood sampling to evaluate the heart's anatomy and function and to obtain samples for subsequent blood-based biomarker analyses.

Additionally, saliva may be sampled and/or neonatal blood samples from national biobank storage will be retrieved for comparison with cardiovascular biomarker profiles in these controls if available.

To evaluate these cardiovascular assessments in predefined age groups, a subgroup of these participating subjects will be asked to complete additional cardiac magnetic resonance imaging based on study protocols.

Incidental findings of congenital heart disease will be followed up according to standard care protocols in designated paediatric cardiology clinics throughout the participating healthcare regions in Sweden.

A subgroup of cases with congenital heart disease that lead to pulmonary over-circulation, such as atrial and ventricular septal defects, partial anomalous pulmonary venous drainage, aorto-pulmonary windows and patent ductus arteriosus, will be asked to participate if the lesion has not been treated by open heart surgery or cardiac catheter interventions at enrolment.

Subjects with these predefined types of congenital heart disease aged 0-17 years at enrolment will undergo standard electrocardiograms (ECG), echocardiography and blood sampling to assess biomarkers at baseline and at 6-12 month follow-up intervals in dedicated paediatric cardiology clinics over a maximum period of three years.

Saliva samples and/or cardiovascular tissue obtained during open heart surgery may also be analysed for studied cardiovascular biomarkers. Additionally, neonatal blood samples from national biobank storage will be retrieved for comparison with current biomarker profiles if available.

For those congenital heart disease cases referred for open heart surgery or cardiac catheter intervention to correct the congenital heart lesion based on standard care assessment decisions during the study period, follow-up will end one year after such intervention. To evaluate cardiovascular assessments in predefined age groups, a subgroup of participating cases will be asked to complete additional cardiac magnetic resonance imaging based on study protocols.

Prospective evaluation of developed blood-based biomarkers assays and novel cardiac imaging biomarkers of heart function in infants and children will be further assessed to evaluate the feasibility of these methods to timely and precisely identify newborns with congenital heart disease by combined blood-based biomarker analyses and to assess whether newly identified functional parameters on heart function would be suitable to guide clinical risk-assessment and decision-making processes in terms of type and timing of cardiac interventions . These imaging biomarkers will, for example, evaluate the usefulness of measuring kinetic energy within the left ventricle of the heart in children with congenital heart disease based on magnetic resonance and echocardiography methods.

ELIGIBILITY:
Inclusion Criteria:

* obtained written informed consent prior to enrolment
* resident within participating healthcare regions in Sweden during study
* age 0-17 years at enrolment
* Controls: No evidence of congenital heart disease and no history of cardiovascular disease
* Cases: congenital heart lesions prior to open heart surgery or cardiac catheter intervention with grouping into i.e. ventricular septal defects and atrial septal defects, complex and critical cases requiring infant surgery or patency of the arterial duct to maintain the circulation postnatally.

Exclusion Criteria:

* inability to obtain written informed consent prior to study enrolment and/or comply with study protocol
* non-resident in participating healthcare regions of Sweden during study
* age more than 17 years at enrolment
* presence of congenital heart disease where the lesion has already been treated by open heart surgery or cardiac catheter intervention
* participation in other research study with conflicting aims / interests

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Time from diagnosis to open-heart surgery or cardiac catheter intervention in predefined congenital heart disease lesions | 3 years
  Number of days from date of diagnosis of predefined congenital heart disease lesion until date of open-heart surgery or cardiac catheter intervention to treat lesion

SECONDARY OUTCOMES:
Screening for congenital heart disease in newborns using circulating biomarkers in blood samples | 3 years
  Results will be based on circulating biomarker analysis in infants using dried blood spot samples to improve detection of congenital heart disease. Results in normal controls will be compared to predefined congenital heart disease lesions and results expressed in ng/l using cardiovascular biomarkers such as NT-proBNP and IL1RL1 (ST2).
Circulating cardiovascular protein biomarker profiling in infants and children with predefined congenital heart disease lesions vs normal controls using blood samples. | 3 years
  Circulating biomarker profiling results will be expressed in 'NPX' units (Normalized Protein eXpression concentrations from proximity extension assay analyses of protein concentrations in blood samples using O-link's 'Target 96 cardiovascular III' panel, link: https://www.olink.com/products/cvd-iii-panel/)
Measurement of cardiac magnetic resonance 4-dimensional flows to estimate 'kinetic energy' supported by advanced echocardiography in normal controls vs predefined lesions of congenital heart disease | 3 years
  Results will be based on cardiac magnetic resonance 4D flow and supported by advanced echocardiographic assessments and expressed as kinetic energy (milli Joule) to assess for normal and abnormal patterns of cardiac function.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Clausen, MD, Principal Investigator — Children's Heart Centre, University Hospital of Lund
Locations (1):
- Children's Heart Centre at Lund's University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymised clinical data relevant to the publication process of peer-reviewed scientific journals may be made available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 2024
Access Criteria: After conclusion of the study, anonymised clinical data may be may available after reasonable request to medical researcher in recognised non-profit academic institutions

DOCUMENTS (3):
  • Study Protocol (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04667455/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04667455/SAP_001.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04667455/ICF_002.pdf